CLINICAL TRIAL: NCT06798948
Title: Effect of the Combined Application of Cynara Scolymus, Silybum Marianum, Curcuma Longa, and Glycyrrhiza Glabra in Improving Metabolic Associated Fatty Liver Disease : a Randomized Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Lab,MD (Other Government)
Collaborators: Xin Hua Hospital of Zhejiang Province (Other)
Responsible Party: Sponsor-Investigator, Li Lab,MD, Prof., Zhejiang Chinese Medical University
Organization: Zhejiang Chinese Medical University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Evaluation of CSCG on MAFLD
Record Dates: First submitted 2025-01-14; First posted 2025-01-29 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Metabolic-associated Fatty Liver Disease (MAFLD)
Keywords: Metabolic-associated fatty liver disease (MAFLD); MRI-PDFF; Chinese Medcine
MeSH Terms: interventions — milk-thistle extract; turmeric extract; Glycyrrhiza glabra extract

STUDY DESIGN:
Intervention Model Description: Intervention Group: combination of cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra Control Group: placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra (Experimental): The patient takes two tablets of the mixture cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra every day.
  Interventions: Dietary Supplement: Combination of cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra
- maltodextrin group (Placebo Comparator): The patient takes two tablets of the placebo maltodextrin every day
  Interventions: Other: Placebo maltodextrin

INTERVENTIONS:
Dietary Supplement: Combination of cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra — Oral combination of cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra
  Arms: Combination of cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra
Other: Placebo maltodextrin — The patient takes two tablets of the placebo maltodextrin every day
  Arms: maltodextrin group

SUMMARY:
Metabolic-associated fatty liver disease (MAFLD) is a chronic progressive liver disease caused by nutrient excess and insulin resistance (IR) in genetically susceptible individuals. With the prevalence of obesity and type 2 diabetes, the morbidity and incidence of MAFLD have been increasing globally, particularly in China. MAFLD and metabolic syndrome as well as type 2 diabetes are mutually causal, jointly promoting the incidence of atherosclerotic cardiovascular disease, chronic kidney disease, liver decompensation, and malignant tumors such as hepatocellular carcinoma. MAFLD has become an increasingly severe public health issue in China. Effective clinical interventions for MAFLD patients are of great public health significance for the prevention of terminal diseases.

Cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra are traditional Chinese medicinal herbs that have demonstrated significant effectiveness in improving metabolic diseases. Cynara scolymus contains polyphenols, flavonoids, terpenes, and other substances, possessing antioxidant, anti-aging, anti-tumor, anti-microbial, antihypertensive, and kidney-tonifying properties. Silybum marianum belongs to the Compositae family and has the effects of clearing heat and detoxifying, soothing the liver, and promoting bile flow. The active ingredient of silybum marianum is silymarin, a flavonoid compound, which has antioxidant and anti-hepatic fibrotic effects, protecting hepatocytes from damage by free radicals and promoting hepatocyte regeneration and repair. Curcuma longa is a flowering plant of the zingiberaceae family, and its active ingredient curcumin has multiple functional properties such as anti-tumor, anti-inflammatory, hypoglycemic, and antioxidant activities. Glycyrrhiza glabra is one of the commonly used medicinal plants, possessing the effects of clearing heat and detoxifying, tonifying the spleen and benefiting qi, nourishing the lungs, and resolving phlegm. Its main active ingredients include triterpenoid saponins, flavonoids, and polysaccharides, which exhibit various pharmacological effects such as antioxidant, immunoregulatory, antiviral, and anti-tumor activities. At the human population level, there is currently no research on the combined intervention of cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra in patients with MAFLD.

Therefore, this study intends to conduct a randomized controlled double-blind trial to explore the effects of the combined application of cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra on liver function, liver fat content, glucose and lipid metabolism, and other aspects in patients with MAFLD, in order to clarify the health improvement effects of this combined intervention in patients with MAFLD and provide population-based evidence and strategies for health promotion in this patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who meet the clinical diagnostic criteria for metabolic-associated fatty liver disease and have mild to moderate fatty liver.
2. Aged 18-65, regardless of gender.
3. Have not taken any liver-protecting medications in the past 3 months.
4. Informed subjects who voluntarily sign the informed consent form and agree to participate in all visits and treatments as required by the trial protocol.

Exclusion Criteria:

1. Excessive alcohol consumption or inability to quantify alcohol consumption within the past 12 months (weekly ethanol intake: ≥210g for males, ≥140g for females).
2. Currently pregnant and/or lactating women, or women planning to become pregnant within the next 3 months.
3. Diagnosed with allergies or other known or suspected allergic reactions (systemic, inhaled, or localized), with a history of sensitivity to ingredients in the product formula.
4. Previous or current use of liver-protecting products containing ingredients such as cynara scolymus, silybum marianum, curcuma longa, and glycyrrhiza glabra , etc.
5. Coexisting with other hepatobiliary diseases, such as autoimmune liver disease, viral hepatitis, liver fibrosis, cirrhosis, drug-induced liver disease, Wilson's disease, etc.
6. Diagnosed with obesity, hypertension, and/or diabetes and taking relevant therapeutic drugs (e.g., orlistat for obesity treatment, statins for lipid-lowering, hydrochlorothiazide, metoprolol, bisoprolol for hypertension treatment, metformin, dapagliflozin for diabetes treatment, etc.).
7. Coexisting with specific diseases that can lead to fatty liver, such as total parenteral nutrition, abetalipoproteinemia, congenital lipoatrophic diabetes, celiac disease, etc.
8. Long-term use of drugs known to cause hepatic steatosis or steatohepatitis (e.g., amiodarone, methotrexate, tamoxifen, glucocorticoids, etc.).
9. Coexisting with severe cardiovascular and cerebrovascular diseases or renal insufficiency.
10. Unstable weight and metabolic parameters within 6 to 8 weeks before randomization, with weight changes exceeding 5% or rapid weight loss (>1.6 kg/week).
11. History of malignancy within the past five years (except for localized skin basal cell carcinoma), regardless of recurrence or metastasis.
12. History of immunosuppression or immunodeficiency disorders (including HIV or AIDS), or current use of immunosuppressive drugs or radiotherapy.
13. Chronic diseases and endocrine disorders such as asthma, epilepsy, hyperthyroidism or hypothyroidism, and/or the use of corresponding therapeutic drugs.
14. History of drug abuse.
15. History of antibiotic use within the past month.
16. Participation in other population intervention studies within the past 3 months or receipt of other non-study group treatments during the study.
17. Other conditions or diseases that, in the judgment of other researchers, may reduce the likelihood of enrollment or complicate the enrollment process, such as frequent changes in work environment, unstable living environment, etc., which may lead to loss to follow-up; inconvenience in daily living, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging proton density fat fraction in hepatic steatosis | Baseline, up to 12 weeks of the study
  Magnetic Resonance Imaging (MRI) technology utilizes magnetic fields and radiofrequency pulses to conduct non-invasive examinations of tissues. When measuring liver fat content, MRI employs water-fat separation techniques to quantify the proton density of water molecules and fat molecules (PDFF) within the liver, thereby providing a quantitative analysis of fat content.

SECONDARY OUTCOMES:
Liver function | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  Alanine aminotransferase (ALT), aspartate aminotransferase (AST), γ-glutamyltransferase (γ-GT), alkaline phosphatase (ALP), total bilirubin (TBIL), direct bilirubin (DBIL), indirect bilirubin (IBIL), alcohol dehydrogenase (ADH), aldehyde dehydrogenase (ALDH)
Glucose metabolism | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  Hemoglobin A1c (HbA1c)
Glucose metabolism | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  Fasting blood glucose
Lipid metabolism | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  Serum triglycerides (TG), total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), apolipoprotein A-I (ApoA-I), apolipoprotein B (Apo B).

OTHER OUTCOMES:
Inflammation level | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  High-sensitivity C-reactive protein (hs-CRP)
Inflammation level | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  tumor necrosis factor (TNF-α)
Inflammation level | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  interleukins (IL-1β, IL-6).
Intestinal flora | Baseline, up to 12 weeks of the study
  16s rRNA sequencing
Kidney function | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  Blood creatinine (CREA), urea nitrogen (BUN), uric acid (UA)
Blood routine test | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  Blood routine examination indicators
Urine Routine Test: | Baseline, up to 6 weeks， up to 12 weeks，up to 16 weeks of the study
  Urinalysis examination indicators

CONTACTS AND LOCATIONS:
Overall Officials: Songtao Li, Study Chair — Zhejiang Chinese Medical University
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Select...
  - Zhejiang Xinhua Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Protect volunteers' personal health data and personal privacy

REFERENCES:
- [Background] Li BY, Xi Y, Liu YP, Wang D, Wang C, Chen CG, Fang XH, Li ZX, Chen YM. Effects of Silybum marianum, Pueraria lobate, combined with Salvia miltiorrhiza tablets on non-alcoholic fatty liver disease in adults: A triple-blind, randomized, placebo-controlled clinical trial. Clin Nutr ESPEN. 2024 Oct;63:2-12. doi: 10.1016/j.clnesp.2024.06.003. Epub 2024 Jun 10. PMID 38879879
- [Background] Wang X, Jin Y, Di C, Zeng Y, Zhou Y, Chen Y, Pan Z, Li Z, Ling W. Supplementation of Silymarin Alone or in Combination with Salvianolic Acids B and Puerarin Regulates Gut Microbiota and Its Metabolism to Improve High-Fat Diet-Induced NAFLD in Mice. Nutrients. 2024 Apr 14;16(8):1169. doi: 10.3390/nu16081169. PMID 38674860
- [Background] Hansen CD, Gram-Kampmann EM, Hansen JK, Hugger MB, Madsen BS, Jensen JM, Olesen S, Torp N, Rasmussen DN, Kjaergaard M, Johansen S, Lindvig KP, Andersen P, Thorhauge KH, Brond JC, Hermann P, Beck-Nielsen H, Detlefsen S, Hansen T, Hojlund K, Thiele MS, Israelsen M, Krag A. Effect of Calorie-Unrestricted Low-Carbohydrate, High-Fat Diet Versus High-Carbohydrate, Low-Fat Diet on Type 2 Diabetes and Nonalcoholic Fatty Liver Disease : A Randomized Controlled Trial. Ann Intern Med. 2023 Jan;176(1):10-21. doi: 10.7326/M22-1787. Epub 2022 Dec 13. PMID 36508737
- [Background] Dellinger RW, Holmes HE, Hu-Seliger T, Butt RW, Harrison SA, Mozaffarian D, Chen O, Guarente L. Nicotinamide riboside and pterostilbene reduces markers of hepatic inflammation in NAFLD: A double-blind, placebo-controlled clinical trial. Hepatology. 2023 Sep 1;78(3):863-877. doi: 10.1002/hep.32778. Epub 2022 Nov 22. PMID 36082508